CLINICAL TRIAL: NCT02169882
Title: A Randomized Double Blinded Phase 2b Clinical Trial Comparing Standard Dose With Two Higher Doses of Rifampicin for Treatment of Adults With Tuberculous Meningitis
Brief Title: High-dose Rifampicin for the Treatment of Tuberculous Meningitis: a Dose-finding Study
Acronym: ReDEFINe
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TB-201406.01; PGA-2000003601 (Other: PEER Health)
Record Dates: First submitted 2014-06-15; First posted 2014-06-23 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2016-12

CONDITIONS: Tuberculosis, Meningeal
Keywords: Tuberculous meningitis; Rifampicin; Dose finding study; Pharmacokinetics
MeSH Terms: conditions — Tuberculosis, Meningeal | interventions — Rifampin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rifampicin 450 mg (standard dose) (Active Comparator): Twenty patients will receive 1 tablet of 450 mg Rifampicin and 2 tablets of placebo once daily for 30 days.
  Unconscious subjects will receive oral drugs via nasogastric tubes (NGT).
  After completion of one-month treatment, patients will receive 1 tablet of 450 mg Rifampicin.
  Along with study drug and placebo, patients will receive other oral TB drugs (INH, Ethambutol, and Pyrazinamide) and pyridoxin, in accordance to National TB Program guidelines for 6 months.
  Patients will also receive dexamethasone in decreasing dose (in 6-8 weeks, according to TBM severity grade on admission)
  Interventions: Drug: Placebo; Drug: Other TB drugs; Drug: Adjuvant dexamethasone
- Rifampicin 900 mg per oral (Experimental): Twenty patients will receive 2 tablets of 450 mg Rifampicin and 1 tablet of placebo once daily for 30 days.
  Unconscious subjects will receive oral drugs via nasogastric tubes (NGT)
  After completion of one-month treatment, patients will receive 1 tablet of 450 mg Rifampicin.
  Along with study drug and placebo, patients will receive other oral TB drugs (INH, Ethambutol, and Pyrazinamide) and pyridoxin, in accordance to National TB Program guidelines for 6 months.
  Patients will also receive dexamethasone in decreasing dose (in 6-8 weeks, according to TBM severity grade on admission)
  Interventions: Drug: Placebo; Drug: Rifampicin; Drug: Other TB drugs; Drug: Adjuvant dexamethasone
- Rifampicin 1350 mg per oral (Experimental): Twenty patients will receive 3 tablets of 450 mg Rifampicin and 0 tablet of placebo once daily for 30 days.
  Unconscious subjects will receive oral drugs via nasogastric tubes (NGT)
  After completion of one-month treatment, patients will receive 1 tablet of 450 mg Rifampicin.
  Along with study drug and placebo, patients will receive other oral TB drugs (INH, Ethambutol, and Pyrazinamide) and pyridoxin, in accordance to National TB Program guidelines for 6 months.
  Patients will also receive dexamethasone in decreasing dose (in 6-8 weeks, according to TBM severity grade on admission)
  Interventions: Drug: Rifampicin; Drug: Other TB drugs; Drug: Adjuvant dexamethasone

INTERVENTIONS:
Drug: Placebo — Patients receiving 450 mg rifampicin will receive additional 2 placebo tablets, while those who receive 900 mg rifampicin will receive 1 placebo tablet.
  Patients receiving 1350 mg rifampicin will not receive any placebo tablet.
  With this arrangement, every subject will receive 3 tablets of study drugs.
  Arms: Rifampicin 450 mg (standard dose); Rifampicin 900 mg per oral
Drug: Rifampicin — Patients in experimental arms will receive either 1 or 2 additional tablets of rifampicin.
  Placebo tablets will be added accordingly, so that every study subject will receive 3 tablets of rifampicin plus placebo as described in the Arms section.
  Other Names: Rifampisin - Kimia Farma
  Arms: Rifampicin 1350 mg per oral; Rifampicin 900 mg per oral
Drug: Other TB drugs — Along with study drug and placebo, patients will receive other oral TB drugs (INH, Ethambutol, and Pyrazinamide) and pyridoxin, in accordance to National TB Program guidelines for 6 months.
  Unconscious subjects will receive oral drugs via nasogastric tubes (NGT)
Drug: Adjuvant dexamethasone — Patients will receive dexamethasone in decreasing dose (in 6-8 weeks, according to TBM severity grade on admission)

SUMMARY:
Tuberculous meningitis (TBM) is the most severe form of tuberculosis infection with high mortality. Current treatment regimens are not based on clinical trials. Rifampicin is a key drug for TBM, but its penetration into the brain is limited, suggesting that a higher dose may be more effective.

There are several highly relevant, outstanding questions related to the appropriate dose of rifampicin for TBM, before a multicenter phase 3 trial can be performed. These are:

1. Previous phase 2a randomized clinical trial (done in the same setting as this proposed study) suggests that high doses of intravenous rifampicin (600mg, circa 13 mg/mg) for TBM is safe and associated with a survival benefit in adults. Given that i.v. rifampicin is not readily available, this needs to be confirmed using an equivalent higher oral dose of rifampicin.
2. Recent pharmacokinetic analysis of a continuation trial comparing 600 mg i.v. rifampicin with 750 mg and 900 mg oral rifampicin suggests that an even higher dose may be needed; but this has not been examined
3. Based on those previous data, there is a need to explore a longer duration of high-dose rifampicin for a subsequent phase 3 randomized clinical trial; treatment response in the investigators previous trial suggest that the optimal duration may be > 14 days.
4. There is a need to explore relevant treatment endpoints besides mortality including neurological, neuroradiological and inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, aged 15 years or above.
2. Clinical suspicion of TBM and CSF/blood glucose ratio < 0.5.
3. None or less than 3 days of anti-tuberculosis chemotherapy taken for the current infection.
4. Patient or representative (if the patient is incapacitated) is willing and able to give informed consent for participation in the study.
5. Willingness to allow storage of specimens.

Exclusion Criteria:

Patients may not enter the study if any of the following apply:

1. Liver dysfunction (ALT > 5 times upper limit); kidney dysfunction (eGFR < 50 ml/min)
2. Pregnancy or breastfeeding (negative urine pregnancy test for all females of child-bearing age).
3. Confirmed cryptococcus meningitis (LFA), or confirmed bacterial meningitis (microscopy).
4. Rapid clinical deterioration at time of presentation (e.g. signs of sepsis, decreasing consciousness or signs of cerebral oedema, or herniation)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2016-11-05 (Actual); Study Completion 2017-05-05 (Actual)

PRIMARY OUTCOMES:
Rifampicin concentrations in plasma and cerebrospinal fluid (CSF) | Day 2 (+/- 1) after administration of study drugs
  The rifampicin concentrations in plasma are measured from blood samples that are obtained by intensive pharmacokinetic sampling at 6 sampling time points (h0, 1, 2, 4, 8, 12 post dose). CSF rifampicin concentration will be measured using CSF sample taken by means of lumbar puncture at hour 3-6 post dose at the same day of blood sampling.

SECONDARY OUTCOMES:
Rifampicin concentrations in plasma and CSF at steady-state | Day 10 (+/- 1) after starting treatment with study drugs
  The rifampicin concentrations in plasma are measured from blood samples that are obtained by intensive pharmacokinetic sampling at 6 sampling time points (h0, 1, 2, 4, 8, 12 post dose). CSF rifampicin concentration will be measured using CSF sample taken by means of lumbar puncture at hour 3-6 post dose at the same day of blood sampling.
Grade 3 and 4 and serious adverse events | Within 60 days
  Determined by measurement of liver function, hematology, gastrointestinal intolerance and hypersensitivity at days 3, 7, 10, 14, 30, 45, and 60
Mortality | 180 days
Neurological response | Within 60 days
  Neurological responses that show both improvement (e.g. time to resolution of comma, time to fever resolution) and worsening (time to development of neurological deficits) will be measured and recorded at days 3, 7, 30 and 60.
Neuroradiological response | 60 days
  Development of infarction or other complication of TBM will documented by performing and comparing brain MRIs that will be done within the first 5 day and 60 day (+/- 5 days) after randomization
Resolution of blood and CSF inflammatory response | 7 days
  Inflammatory response will be measured at day 0 and day 7
Sensitivity of GeneXpert for diagnosing TBM | Within 6 weeks
  Every CSF sample from patients who come with suspicion of TBM will be inoculated in GeneXpert cartridge and standard culture measures (MODS), and the result will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Rovina Ruslami, M.D., PhD, Principal Investigator — Faculty of Medicine Universitas Padjadjaran, Bandung, Indonesia
Locations (1):
- Hasan Sadikin General Hospital, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruslami R, Ganiem AR, Dian S, Apriani L, Achmad TH, van der Ven AJ, Borm G, Aarnoutse RE, van Crevel R. Intensified regimen containing rifampicin and moxifloxacin for tuberculous meningitis: an open-label, randomised controlled phase 2 trial. Lancet Infect Dis. 2013 Jan;13(1):27-35. doi: 10.1016/S1473-3099(12)70264-5. Epub 2012 Oct 25. PMID 23103177
- [Derived] Dian S, Yunivita V, Ganiem AR, Pramaesya T, Chaidir L, Wahyudi K, Achmad TH, Colbers A, Te Brake L, van Crevel R, Ruslami R, Aarnoutse R. Double-Blind, Randomized, Placebo-Controlled Phase II Dose-Finding Study To Evaluate High-Dose Rifampin for Tuberculous Meningitis. Antimicrob Agents Chemother. 2018 Nov 26;62(12):e01014-18. doi: 10.1128/AAC.01014-18. Print 2018 Dec. PMID 30224533